CLINICAL TRIAL: NCT01412138
Title: "Identification, Characterization and Isolation of Somatic Stem Cells in Human Endometrium of Women With Endometriosis"
Brief Title: Somatic Stem Cells in Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Carlos Simon, Principal Investigator, Instituto Valenciano de Infertilidad, IVI VALENCIA
Other Study IDs: 1006-C-073-CS-F
Record Dates: First submitted 2011-07-28; First posted 2011-08-09 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Genetic Testing

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrial biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARM 1: ENDOMETRIAL SAMPLE
  Interventions: Other: genetic analysis

INTERVENTIONS:
Other: genetic analysis — 1. To identify by flow cytometry through technique of "Side Population" the population of somatic stem cells present in both human endometrial eutopic and ectopic endometrium of women with ovarian endometriosis, peritoneal and recto-vaginal.
  2. In vitro culture conditions for cell proliferation.
  3. To characterize the somatic stem cell population using techniques of endometriotic cell and molecular biology.
  4. Compare the results obtained from patients with endometriosis with control patients (without endometriosis) earlier work by our group.

SUMMARY:
Human endometrium is a very dynamic tissue characterized by cyclical process of proliferation, differentiation and cellular shedding as part of each menstrual cycle. This issue suggests the presence of somatic stem cells. Endometriosis is characterized by presence of endometrium outside the uterine cavity. The existence of a somatic stem cell population in endometrium could explain the incorrect proliferation of these cells, which would lead to formation of endometriotic foci.

DETAILED DESCRIPTION:
Throughout the life of the woman, the endometrium undergoes a series of continuous modifications that require a highly accurate feedback mechanism and specialized and must be based on the activity of the stem cell population.

Endometriosis is an estrogen-dependent chronic disease characterized by the presence of functional endometrium outside the uterine cavity, mainly in the peritoneum and ovary (Giudice and Kao, 2004). It affects 6-10% of women of reproductive age, often resulting in a series of gynecological problems, including dysmenorrhea, pelvic pain and infertility. The nature of endometriosis suggests that the initiation of ectopic endometrial lesions may be due to stem or progenitor cells, which is consistent with the theory of retrograde menstruation (Starzinski-Powitz et al. 2001; Leyendecker et al. 2002, Gargett, 2006; Gargett, 2007, Sasson and Taylor, 2008). To date, no direct evidence of the role of somatic stem cells of the endometrium in the pathogenesis of endometriosis. However, numerous studies show that ectopic endometrial cells implant in many established models used for the study of endometriosis.(Masuda et al., 2007b; Sasson and Taylor, 2008; Gargett y Masuda.,2010)

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients with endometriosis:

1. Female patients with ovarian endometriosis, peritoneal and recto-vaginal.
2. Aged between 20 and 40.
3. Signing of informed consent for collection and storage of biological samples.

Exclusion Criteria:

1. Contraindications for endometrial biopsy.
2. Failure to sign informed consent for collection and storage of biological samples.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with endometrial infertility factor, undergoing ART.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Characterization of endometrial stem cells through Flow Citometry and Side Population techniques and In vitro culture cellular proliferation to then characterize the cell population through molecular and cellular techniques. | TWO YEARS

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simon, MDPhd, Principal Investigator — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Spain